CLINICAL TRIAL: NCT06102733
Title: Chronic Pelvic Pain Management in Female and Male Adult Patients
Brief Title: Chronic Pelvic Pain in Females and Males
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAne2018 Pelvic Pain WoMen
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Pain Syndrome; Sacroiliac Disorder; Piriformis Syndrome; Sacrococcygeal Disorder; Inguinal Hernia
Keywords: Pelvic pain
MeSH Terms: conditions — Piriformis Muscle Syndrome; Hernia, Inguinal; Pelvic Pain | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult chronic pain patients: Adult chronic pain patients with pelvic, inguinal or sacroiliac pain
  Interventions: Behavioral: Rehabilitation therapy

INTERVENTIONS:
Behavioral: Rehabilitation therapy — Chronic pain rehabilitation therapy

SUMMARY:
Pelvic pain is under-reported in healthy adults. Many patients with pelvic pain under-estimate the problem. Chronic pelvic pain can be managed properly, if diagnosed promptly.

This is a quantitative analysis of prospective clinical data. It evaluates the management of pelvic pain in a cohort population, and analyzes the treatment outcome.

DETAILED DESCRIPTION:
Pelvic pain is common, but under-reported in healthy adults. Pelvic pain is reported more commonly in women than in men. Many patients with pelvic pain under-estimate the severity of the problem. Chronic pelvic pain can be managed successfully, if diagnosed properly. Many combinations of multimodal analgesia and rehabilitation therapy may be safe and effective for pelvic pain.

This study is a quantitative analysis of prospective clinical data. It is an evaluation of the prevalence and management of pelvic pain in a cohort population of chronic pain patients. This is an analysis of multimodal analgesia types, rehabilitation therapy types, treatment outcome, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pelvic pain
* Patients with sacroiliac pain
* Patients with inguinal pain
* Patients with coccygeal pain
* Patients with piriformis pain

Exclusion Criteria:

* Patients with spinal pain
* Patients who had spine surgery

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic pelvic pain who undergo treatment in pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score, objective measurement using the validated Numeric Pain Rating scale | 12 months
  Pain score, using the Numeric Pain Rating scale of 0 to 10, low scores indicate less pain, high scores indicate worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Olumuyiwa Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No